CLINICAL TRIAL: NCT05165576
Title: The Influence of Child-centered Communication on Children's Anxiety and Use of Anesthesia for MRI
Brief Title: Child-centered Communication and Anesthesia Use for MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade do Porto (Other)
Collaborators: Centro Hospitalar De São João, E.P.E. (Other); Centro de Investigação em Tecnologias e Serviços de Saúde (Other); Rede de Investigação em Saúde (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CASTRO
Record Dates: First submitted 2021-11-22; First posted 2021-12-21 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2021-11

CONDITIONS: Behavioral Problem of Child; Anxiety
Keywords: patient-centered communication; children; MRI; anesthesia; toy simulation
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: The investigator applied the intervention. The participant and the outcomes assessors were blind as to which group participants were assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Child-centered communication (Experimental): The child's preparation for the MRI scanning is conducted using a child-centered communication type of interaction
  Interventions: Behavioral: Child-centered communication
- Magnetic Resonance Imaging (MRI) Simulation Toy (Active Comparator): The child's preparation for the MRI scanning is conducted through provision of general information about the MRI exam simulated with an MRI toy
  Interventions: Behavioral: Child-centered communication
- General information about the Magnetic Resonance Imaging (MRI) exam (No Intervention): The child's preparation for the MRI scanning is based on the provision of routine information about the MRI exam

INTERVENTIONS:
Behavioral: Child-centered communication — The child is asked for ideas, fears and concerns regarding the magnetic resonance imaging exam and responses are tailored to these individual needs
  Arms: Child-centered communication; Magnetic Resonance Imaging (MRI) Simulation Toy

SUMMARY:
The goal of this project is to study the influence of child-centered communication on children's anxiety, satisfaction and the use of anesthesia for MRI

DETAILED DESCRIPTION:
This study seeks to inspect the influence of a child-centered communication (CCC) on anesthesia use in magnetic resonance imaging (MRI) exams among four- to 10-year-old children. Children's levels of anxiety and satisfaction with the interaction also are assessed. Children are divided into three groups by order of arrival. Group 1 receives routine information about the MRI and simulates it with an MRI toy (EG1). Group 2 simulates the exam with the toy and receives the CCC. These two groups are compared with a third group of children who had received only the routine information about the exam and who served as a comparison group (CG).

ELIGIBILITY:
Inclusion Criteria:

* Ages between four and 10 years old
* Having a medical request for the MRI in the hospital
* The MRI performed for the first time

Exclusion Criteria:

* Presenting cognitive, psychiatric or neurological conditions that prevented the understanding of communication
* Having any intra-body devices that impeded performance of the MRI exam

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Anesthesia count | 30 minutes (after the Magnetic Resonance Imaging)
  Number of children who perform the Magnetic Resonance Imaging exam using anesthesia

SECONDARY OUTCOMES:
Change in self-reported anxiety | 20 minutes (before and after the child's preparation)
  Change in anxiety levels before and after preparation for the Magnetic Resonance Imaging, assessed through a self-report question responded on a 1 ("very calm") to 5 ("very scared") scale
Change in heart rate frequency | 20 minutes (before and after the child's preparation)
  Change in anxiety levels before and after preparation for the Magnetic Resonance Imaging assessed through heart rate frequency

OTHER OUTCOMES:
Satisfaction measurement | 20 minutes (after child preparation to do the Magnetic Resonance Imaging)
  Children's satisfaction with the interaction they had in preparation for the Magnetic Resonance Imaging, assessed through self-reported, Yes/No questions

CONTACTS AND LOCATIONS:
Overall Officials: Irene P Carvalho, PhD, Principal Investigator — Universidade do Porto
Locations (2):
- Portugal (2):
  - Centro Hospitalar Universitário de São João, Porto
  - Faculty of Medicine of the University of Porto, Porto

IPD SHARING:
Plan to Share IPD: No
Individual participant data are confidential and will be shared only among the research team. Aggregate data can be shared with others only for research purposes and without any identifiers that might compromise the participant's anonimity